CLINICAL TRIAL: NCT06949007
Title: Yoga for Persistent Post-Surgical Pain (PPSP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Dennis Wilson Munoz Vergara, Instructor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2025P001082; 1K01AT012889-01 (NIH)
Record Dates: First submitted 2025-04-14; First posted 2025-04-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Persistent Post-surgical Pain
Keywords: Persistent Post-Surgical Pain; Yoga; Randomized Controlled Trial; Chronic Pain Health Education
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga group (Experimental): Yoga Program Procedure This program was adapted and validated from a previously validated yoga program for patients with chronic lower back pain (cLBP), originally designed and clinically evaluated by Dr. Saper. While the program includes postures targeting the torso, modifications were made to address the specific needs of post-surgical patients (e.g., verbal intensity cues, duration of pose holding, and posture adjustments).
  The adaptation and validation process was guided by a modified Delphi approach with an embedded focus group, involving both an expert panel and PPSP participants. Participants attended a sample yoga class and shared insights during a focus group discussion, which informed program modifications.
  Interventions: Behavioral: Yoga
- Chronic Pain Health Education (CPHE) (Active Comparator): Chronic Pain Health Education Procedures (CPHE) To partially control for attention and expectation effects associated with yoga therapy, participants randomized to the control group will receive a modified version of an education-based intervention that we recently developed and validated for an ongoing study evaluating migraine pain.
  Participants assigned to the CPHE (Chronic Pain Health Education) arm will attend 12 interactive 15-30-minute education sessions delivered via video conference. Each session will be offered three times per week, allowing participants the option to attend multiple sessions to reinforce the material.
  Most sessions will include a short educational video, which will be watched together by participants and the RA. After each video, the RA will facilitate a structured, scripted discussion on the topic. Example session topics include: Understanding Clinical Trials, Biology of Persistent Post-Surgical Pain (PPSP).
  Interventions: Behavioral: Chronic Pain Health Education

INTERVENTIONS:
Behavioral: Yoga — Duration: 12 weeks; Class length: Three ∼75-minute classes per week. Two in-person/virtual (hybrid), one virtual only (MGB Zoom); Frequency: Three classes per week; Group size: 8-9 PPSP patients.
  Other Names: Yoga exercise
  Arms: Yoga group
Behavioral: Chronic Pain Health Education — Duration: 12 weeks (short videos and PowerPoint presentations); Class length: Interactive 15-30 minute education sessions delivered via video conference (i.e., MGB Zoom); Frequency: Three classes per week; Group size: 8-9 PPSP patients.
  Other Names: CPHE
  Arms: Chronic Pain Health Education (CPHE)

SUMMARY:
The overall goal of this project is to complete a pilot feasibility randomized controlled trial (RCT) to inform a future fully-powered translational study evaluating yoga for management and resolution of persistent-post surgical pan (PPSP) and the role of biological, psychophysical, and psychosocial modulators in PPSP resolution.

DETAILED DESCRIPTION:
More than 100 million people in the United States (US) undergo surgical procedures each year. These individuals are at risk of developing persistent post-surgical pain (PPSP), with estimates as high as 70% for some procedures (e.g., post-thoracotomy, hernial repair, cholecystectomy, cesarean section, sternotomy). PPSP, defined as pain in the surgical area that lasts more than 3 months after surgery, is a unique syndrome of chronic pain. Prior studies suggest that inflammation plays a major role in the development of PPSP, along with peripheral and central sensitization due to nerve damage, and weakening of the endogenous central opioid and endocannabinoid systems. Thus, PPSP provides a unique opportunity that invites translational research.

Currently, the main strategy for managing PPSP is pharmacological treatment. However, long-term use of potent analgesics is associated with untoward side effects (e.g., priming to develop PPSP). A growing body of research supports the benefit of mind-body movement therapies (MBMT), such as yoga, in treating chronic pain; however, little attention has been devoted to adapting a yoga program for the specific needs that PPSP patients may face (e.g., range of motion). Moreover, while randomized controlled trials (RCTs) support that yoga alleviates pain, the mechanisms underlying its therapeutic benefits are largely unclear.

Preclinical and clinical studies suggest yoga has the potential to alter systemic levels of inflammatory mediators (i.e., cytokines and oxylipins) via body movement and stretching. Given that inflammatory processes may contribute to more severe and prolonged pain after surgery, yoga practice may mitigate the development of PPSP via the modulation of circulating levels of inflammatory and endocannabinoid mediators, resulting in endogenous analgesia. Evaluation of the links between yoga and post-surgical pain, with modulation of systemic levels of these potential mediators, is a novel area of inquiry, which may inform the practical and safe use of yoga in postoperative patients.

This pilot translational RCT proposes comparing a yoga program versus a chronic pain health education (CPHE) program in individuals with PPSP. This pilot RCT will help collect essential preliminary data to inform a future translational trial evaluating a widely available and adaptable intervention (yoga) for a highly prevalent and debilitating pain condition (PPSP) that impacts multiple dimensions of whole-person health.

Multiple indicators of feasibility and acceptability of the intervention and procedures will be evaluated. Upon enrollment, participants (N=50) will be randomly assigned 1:1 to one of the two treatment groups using a permuted block randomization, with block sizes of 2 and 4 to either the yoga group or the health education control group.

Following the study timeline, participants will be asked to complete three assessments: baseline (T1-prior to randomization), post-intervention (T2- ~ 12 weeks post-T1), and 3 months post-intervention (T3- ~24 weeks post-T1). Each assessment will include blood samples for select outcomes related to inflammation (e.g., cytokines), psychophysical assessment of pain and pain sensitivity test (i.e., Quantitative Sensory Testing), psychosocial patient-centered outcomes (i.e., PROMIS-29), clinical neuropathy (i.e., S-LANSS), and self-patient-reported pain interference and severity (i.e., BPI). Participants in the yoga groups (approximately 3 cohorts of 8-9 participants each) will be asked to provide brief feedback on acceptability of session content via a weekly survey.

This study will allow us to address our primary Aim 1: To design and conduct a pilot feasibility RCT of yoga in individuals with PPSP. This aim has three components: a) To adapt a validated yoga program to individuals with PPSP ; b) To assess multiple indicators of feasibility and acceptability, such as recruitment, retention, adherence, and acceptability and; c) To assess feasibility of collecting PPSP-related outcomes. An secondary exploratory Aim 2 will explore the longitudinal relationship between yoga or an education control group on changes in PPSP-related inflammatory markers (e.g., IL-6) and other known psychophysical (i.e., QST), and psychosocial (e.g., PROMIS-29) modulators of PPSP to further inform our conceptual framework and the design of a larger trial assessing the impact of yoga on PPSP resolution.

ELIGIBILITY:
Inclusion Criteria:

* History of torso surgeries. Examples are thoracotomy, sternotomy, mastectomy and breast implant, open abdominal surgeries, and cesarean section
* Completion of surgery alone or surgery and complementary pharmacological treatment
* Being 18 years of age or older
* 3 months with PPSP and 4/10 in BPI severity (clinically considered a moderate range)
* Access to reliable modes of transportation for study visits and yoga classes
* Confirmed access to and proficiency with use of a smartphone, computer, and/or tablet
* Fluent in English.

Exclusion criteria:

* History of joint replacement, amputation, orthopedic (except thoracotomy and sternotomy), and other non-torso surgeries
* Participants with health conditions that lead to difficulty complying with study protocol (i.e., completion of outcome assessments and participation in yoga or CPHE programs), including: Renal dialysis, cognitive impairment, serious neurological or psychiatric disorders; Unstable cardiovascular disease, metastatic cancer, or serious chronic medical condition; Planned surgery during the intervention period; Chronic inflammatory systemic diseases (e.g., rheumatoid arthritis); Active acute or chronic infections requiring antibiotics; Unmanaged hearing or visual impairment affecting participation in virtual classes; Substance use disorder
* Pregnancy or having the intention to become pregnant within the next six months
* Recent (last 3 months) or concurrent participation in weekly MBMT (e.g., yoga, tai chi, qigong) programs, physical therapy, including massage and chiropractic care, or other non-pharmacological treatment as chronic pain management, such as Mindfulness-Based Stress Reduction (MBSR) or meditation
* Recent interventional pain management, defined as procedures such as corticosteroid injection, trigger point injection, and radiofrequency ablation to the cervical or lumbar region within the past 4 weeks and/or scheduled for interventional pain management procedures within the study timeframe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Acceptability for Aim 1-Enrollment | 36 months
  ≥ 30% of contacted eligible participants will enroll. Assessment Instrument: REDCap report.
Feasibility and Acceptability for Aim 1-Retention rate | 36 months
  ≥65% of randomized participants will attend all study visits and complete all outcome assessments.
  Assessment instrument: REDCap Report of three in-person study visits.
Feasibility and Acceptability for Aim 1-Recruitment rate | 36 months
  Recruitment will be completed within 18 months (2-3 participants/month).
  Assessment instrument: REDCap report.
Feasibility and Acceptability for Aim 1-Adherence to interventions (yoga and CPHE) | 36 months
  ≥75% of randomized participants will adhere to the intervention programs. Target: ≥75% Assessment instrument via Mycap survey-Meeting 75% adherence in the 12-week yoga program requires attending at least one class per week for at least 9 weeks. For home practice, 75% adherence (2+ days/week) corresponds to at least 18 sessions over 12 weeks. Participants can meet this goal by virtually attending additional group classes (up to three per week) or by engaging in 15-30 minutes of home practice, recorded in their weekly MyCap survey. Meeting 75% adherence in the 12-week CPHE program requires attending at least one class per week for at least 9 weeks (attendance to weekly PowerPoint presentation and completeness of weekly MyCap survey on CPHE program satisfaction).
Feasibility and Acceptability for Aim 1-Intervention acceptability (yoga and CPHE) | 36 months
  ≥80% of participants will rate the intervention favorably. Target: ≥80% Assessment instrument via REDCap survey asking participants to rate (0=not at all to 10=very much) enjoyment, convenience, helpfulness, and overall satisfaction after each session and at T2 (post-intervention).
Feasibility and Acceptability for Aim 1-Fidelity | 36 months
  ≥70% adherence to the structured yoga class components in 10% of observed classes.
  Assessment instrument: REDCap Report.
Feasibility and Acceptability for Aim 1-Outcome collection | 36 months
  ≥80% of PPSP-related outcome measures will be collected.
  Assessment instruments: REDCap report for clinical, psychophysical, and biological outcome collection.

SECONDARY OUTCOMES:
Exploratory Aim 2-Effect of treatment assignment on PPSP-related psychosocial modulators of PPSP in the yoga and CPHE groups | 48 months
  Descriptive statistics and exploratory treatment assignment effects on clinical outcomes-Brief Pain Inventory (BPI) scores for pain severity (composite of the four pain items-a mean severity score) and interference (mean of the seven interference items).
  Assess at baseline (T1), 12-week post-intervention (T2), and 12-week follow-up (T3). Higher scores indicate greater pain.
Exploratory Aim 2-Effect of treatment assignment on PPSP-related psychosocial modulators of PPSP in the yoga and CPHE groups | 48 months
  Descriptive statistics and exploratory treatment assignment effects on clinical outcomes-PROMIS-29 T scores for the seven domains (Depression, Anxiety, Physical Function, Pain Interference, Fatigue, Sleep Disturbance, and Ability to Participate in Social Roles and Activities).
  Assess at baseline (T1), 12-week post-intervention (T2), and 12-week follow-up (T3).
  A higher PROMIS T-score represents more of the concept being measured.
Exploratory Aim 2-Effect of treatment assignment on PPSP-related psychosocial modulators of PPSP in the yoga and CPHE groups | 48 months
  Descriptive statistics and exploratory treatment assignment effects on clinical outcomes-S-LANSS score from 7 items to assess neuropathic symptoms and signs (range 0-24).
  Assess at baseline (T1), 12-week post-intervention (T2), and 12-week follow-up (T3).
  Higher scores indicate greater neuropathic symptoms and signs.
Exploratory Aim 2-Effect of treatment assignment on PPSP-related psychophysical modulators of PPSP in the yoga and CPHE groups (Temporal summation of pain-TSP) | 48 months
  Descriptive statistics and exploratory treatment assignment effects on psychophysical outcomes-Brief bedside-adapted Quantitative Sensory Testing (QST): Pinprick applicators (force expressed in Newtons and 3-point ordinal scale: absent, impaired, normal) for TSP. Assess at baseline (T1), 12-week post-intervention (T2), and 12-week follow-up (T3).
Exploratory Aim 2-Effect of treatment assignment on PPSP-related psychophysical modulators of PPSP in the yoga and CPHE groups (Painful After Sensation-PAS) | 48 months
  Descriptive statistics and exploratory treatment assignment effects on psychophysical outcomes-Brief bedside-adapted Quantitative Sensory Testing (QST): Pinprick applicators (force expressed in Newtons and 3-point ordinal scale: absent, impaired, normal) for PAS. Assess at baseline (T1), 12-week post-intervention (T2), and 12-week follow-up (T3).
Exploratory Aim 2-Effect of treatment assignment on PPSP-related psychophysical modulators of PPSP in the yoga and CPHE groups (Pressure Pain Threshold-PPTh) | 48 months
  Descriptive statistics and exploratory treatment assignment effects on psychophysical outcomes-Brief bedside-adapted Quantitative Sensory Testing (QST): Algometer (force expressed in units of kilopascals (kPa) or kg/cm2) for PPTh. Assess at baseline (T1), 12-week post-intervention (T2), and 12-week follow-up (T3).
Exploratory Aim 2-Effect of treatment assignment on PPSP-related psychophysical modulators of PPSP in the yoga and CPHE groups (Pressure Pain Tolerance-PPTo) | 48 months
  Descriptive statistics and exploratory treatment assignment effects on psychophysical outcomes-Brief bedside-adapted Quantitative Sensory Testing (QST): Algometer (force expressed in units of kilopascals (kPa) or kg/cm2) for PPTo. Assess at baseline (T1), 12-week post-intervention (T2), and 12-week follow-up (T3).
Exploratory Aim 2-Effect of treatment assignment on PPSP-related biological modulators of PPSP in the yoga and CPHE groups | 48 months
  Descriptive statistics and exploratory treatment assignment effects on inflammatory and analgesic mediators: Multi-analyte flow assay (e.g., customized Legendplex) for cytokines (ng or pg/mL). Lipid extraction and LC-MS-MS or ELISA for oxylipins and endocannabinoids (ng or pg/mL).
  Assess at baseline (T1), 12-week post-intervention (T2), and 12-week follow-up (T3).

CONTACTS AND LOCATIONS:
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
As this pilot study is a randomized trial, unblinded data involving the randomized treatments will be shared after the study database is locked and the main trial findings are disseminated. As done with other trials in the Division of Preventive Medicine at Mass General Brigham, new research collaborations will be encouraged to use the data collected during this trial. Investigators interested in using data from this trial will be directed to contact the principal investigators for data access.
  At all times, we are fully cognizant of and will scrupulously followthe guidelines of the Health Insurance Portability andAccountability Act (HIPAA), to ensure that participants' rights andconfidentiality are not compromised.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Access Criteria: In year 3, data collection and analysis will be completed for dissemination via scientific poster and oral presentations and manuscript publication in peer-reviewed journals.
  In addition, de-identified raw data will be available for up to 5 years at data repositories hosted at the Mass General Brigham Division of Preventive Medicine.
  Findings emanating from this project will be shared principally through manuscripts and oral presentations. Results will be disseminated to physicians and other health practitioners through presentations at scientific meetings and by peer-reviewed manuscript publications in medical and research journals. Furthermore, we will post our results on clinicaltrials.gov.

REFERENCES:
- [Background] Osypiuk K, Ligibel J, Giobbie-Hurder A, Vergara-Diaz G, Bonato P, Quinn R, Ng W, Wayne PM. Qigong Mind-Body Exercise as a Biopsychosocial Therapy for Persistent Post-Surgical Pain in Breast Cancer: A Pilot Study. Integr Cancer Ther. 2020 Jan-Dec;19:1534735419893766. doi: 10.1177/1534735419893766. PMID 32009481
- [Background] Munoz-Vergara D, Grabowska W, Yeh GY, Khalsa SB, Schreiber KL, Huang CA, Zavacki AM, Wayne PM. A systematic review of in vivo stretching regimens on inflammation and its relevance to translational yoga research. PLoS One. 2022 Jun 1;17(6):e0269300. doi: 10.1371/journal.pone.0269300. eCollection 2022. PMID 35648793
- [Background] Berrueta L, Bergholz J, Munoz D, Muskaj I, Badger GJ, Shukla A, Kim HJ, Zhao JJ, Langevin HM. Stretching Reduces Tumor Growth in a Mouse Breast Cancer Model. Sci Rep. 2018 May 18;8(1):7864. doi: 10.1038/s41598-018-26198-7. PMID 29777149
- [Background] Berrueta L, Munoz-Vergara D, Martin D, Thompson R, Sansbury BE, Spite M, Badger GJ, Langevin HM. Effect of stretching on inflammation in a subcutaneous carrageenan mouse model analyzed at single-cell resolution. J Cell Physiol. 2023 Dec;238(12):2778-2793. doi: 10.1002/jcp.31133. Epub 2023 Nov 1. PMID 37909412
- [Background] Schreiber KL, Zinboonyahgoon N, Flowers KM, Hruschak V, Fields KG, Patton ME, Schwartz E, Azizoddin D, Soens M, King T, Partridge A, Pusic A, Golshan M, Edwards RR. Prediction of Persistent Pain Severity and Impact 12 Months After Breast Surgery Using Comprehensive Preoperative Assessment of Biopsychosocial Pain Modulators. Ann Surg Oncol. 2021 Sep;28(9):5015-5038. doi: 10.1245/s10434-020-09479-2. Epub 2021 Jan 15. PMID 33452600
- [Background] Schreiber KL, Martel MO, Shnol H, Shaffer JR, Greco C, Viray N, Taylor LN, McLaughlin M, Brufsky A, Ahrendt G, Bovbjerg D, Edwards RR, Belfer I. Persistent pain in postmastectomy patients: comparison of psychophysical, medical, surgical, and psychosocial characteristics between patients with and without pain. Pain. 2013 May;154(5):660-668. doi: 10.1016/j.pain.2012.11.015. Epub 2012 Dec 5. PMID 23290256
- [Background] Saper RB, Boah AR, Keosaian J, Cerrada C, Weinberg J, Sherman KJ. Comparing Once- versus Twice-Weekly Yoga Classes for Chronic Low Back Pain in Predominantly Low Income Minorities: A Randomized Dosing Trial. Evid Based Complement Alternat Med. 2013;2013:658030. doi: 10.1155/2013/658030. Epub 2013 Jun 26. PMID 23878604
- [Background] Munoz-Vergara D, Rist PM, Yang E, Yeh GY, Lee N, Wayne PM. Oxylipin Dynamics Following A Single Bout of Yoga Exercise: A Pilot Randomized Controlled Trial Secondary Analysis. J Integr Complement Med. 2024 Sep;30(9):897-901. doi: 10.1089/jicm.2024.0233. Epub 2024 Jul 15. PMID 39007170
- [Background] Munoz-Vergara D, Schreiber KL, Langevin H, Yeh GY, Zhu Y, Rist P, Wayne PM. The Effects of a Single Bout of High- or Moderate-Intensity Yoga Exercise on Circulating Inflammatory Mediators: A Pilot Feasibility Study. Glob Adv Health Med. 2022 Dec 11;11:2164957X221145876. doi: 10.1177/2164957X221145876. eCollection 2022. PMID 36583069
- [Background] Saper RB, Lemaster C, Delitto A, Sherman KJ, Herman PM, Sadikova E, Stevans J, Keosaian JE, Cerrada CJ, Femia AL, Roseen EJ, Gardiner P, Gergen Barnett K, Faulkner C, Weinberg J. Yoga, Physical Therapy, or Education for Chronic Low Back Pain: A Randomized Noninferiority Trial. Ann Intern Med. 2017 Jul 18;167(2):85-94. doi: 10.7326/M16-2579. Epub 2017 Jun 20. PMID 28631003
- [Background] Muñoz-Vergara D, Burton W, Bain P, et al. Understanding the dynamics of inflammatory mediators in response to mind-body movement therapies (MBMTs): A systematic review and meta-analysis of studies in healthy subjects. Brain Behavior and Immunity Integrative. 2023;2doi:10.1016/j.bbii.2023.100006
- [Background] Austin PJ, Moalem-Taylor G. The neuro-immune balance in neuropathic pain: involvement of inflammatory immune cells, immune-like glial cells and cytokines. J Neuroimmunol. 2010 Dec 15;229(1-2):26-50. doi: 10.1016/j.jneuroim.2010.08.013. Epub 2010 Sep 25. PMID 20870295
- [Background] Osypiuk K, Kilgore K, Ligibel J, Vergara-Diaz G, Bonato P, Wayne PM. "Making Peace with Our Bodies": A Qualitative Analysis of Breast Cancer Survivors' Experiences with Qigong Mind-Body Exercise. J Altern Complement Med. 2020 Sep;26(9):825-832. doi: 10.1089/acm.2019.0406. PMID 32924562
- [Background] Bower JE, Irwin MR. Mind-body therapies and control of inflammatory biology: A descriptive review. Brain Behav Immun. 2016 Jan;51:1-11. doi: 10.1016/j.bbi.2015.06.012. Epub 2015 Jun 23. PMID 26116436
- [Background] Chapman CR, Vierck CJ. The Transition of Acute Postoperative Pain to Chronic Pain: An Integrative Overview of Research on Mechanisms. J Pain. 2017 Apr;18(4):359.e1-359.e38. doi: 10.1016/j.jpain.2016.11.004. Epub 2016 Nov 28. PMID 27908839